CLINICAL TRIAL: NCT05433727
Title: Dermoscopic Findings of Small Plaque Parapsoriasis and Patch Stage Mycosis Fungoides, Histopathological Correlation With the Dermoscopic Findings and Diagnostic Accuracy of Dermatologists Using Dermoscopic Findings
Brief Title: Dermoscopic Findings of Small Plaque Parapsoriasis and Patch Stage Mycosis Fungoides and Histopathological Correlation
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dilara İlhan Erdil, medical doctor (resident), Istanbul Training and Research Hospital
Other Study IDs: 11.02.2022 karar no:48
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Mycosis Fungoides of Skin
Keywords: mycosis fungoides, parapsoriasis, videodermoscopy
MeSH Terms: conditions — Mycosis Fungoides; Parapsoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — Skin punch biopsy samples routinely taken for diagnostic purposes and which are compatible with mycosis fungoides or parapsoriasis will be evaluated by the pathologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mycosis fungoides group: Patients who routinely have punch skin biopsy for diagnostic purposes and who were both clinically and histopathologically diagnosed with mycosis fungoides will be included. Patients who only have mycosis fungoides patch lesion on their body, over the age of 18, and who have not received topical treatment for the last 2 weeks or systemic therapy for 4 weeks will be included. Demographic, clinical, videodermoscopy, capillaroscopy (lesional) and histopathological data will be recorded.
  Interventions: Diagnostic Test: videodermoscopy, lesional capillaroscopy
- Parapsoriasis group: Patients who routinely have punch skin biopsy for diagnostic purposes and who were both clinically and histopathologically diagnosed with parapsoriasis will be included. Patients who only have parapsoriasis patch lesion on their body, over the age of 18, and who have not received topical treatment for the last 2 weeks or systemic therapy for 4 weeks will be included. Demographic, clinical, videodermoscopy,capillaroscopy (lesional) and histopathological data will be recorded.
  Interventions: Diagnostic Test: videodermoscopy, lesional capillaroscopy

INTERVENTIONS:
Diagnostic Test: videodermoscopy, lesional capillaroscopy — videodermoscopy and lesional capillaroscopy will be performed under different magnification levels to the skin lesions and data will be recorded.

SUMMARY:
Dermoscopic findings of small plaque parapsoriasis and patch stage mycosis fungoides (MF),histopathological correlation of the dermoscopic findings, and using these findings to differentiate two diseases by demonstrating the difference in diagnostic success of dermatologists

DETAILED DESCRIPTION:
Limited number of studies have been conducted on the dermoscopic findings of mycosis fungoides (MF) and small plaque parapsoriasis for the differentiation of these two diseases. Therefore, prospective studies involving a large number of patients and which can reach high magnification levels with videodermoscopy are needed to determine the criteria for discrimination. In our study, dermoscopic demonstration of vascularity will be achieved through videodermoscopy and capillaroscopy from the lesional skin, resulting in high magnification levels (x200).

In terms of histopathology and dermoscopy correlation, skin punch biopsy will be taken for diagnostic purposes. Videodermoscopy and lesional capillaroscopy will be performed to the same site of the lesion where punch biopsy will be taken. As a result patients who had the diagnosis of mycosis fungoides or parapsoriasis will be included to our study. After histopathological features are evaluated by pathologists, dermoscopic correlations will be examined for each lesion.

30 patients with clinical and histopathological diagnosis of mycosis fungoides, and 30 patients with clinical and histopathological diagnosis of small plaque parapsoriasis, who applied to the dermatology clinic of our hospital between february 2022 and june 2022 are included in the study. Patients did not use systemic treatment for 4 weeks and topical treatments in the last 2 weeks were included to the study.

Patient's demographical data, clinical data, videodermoscopy findings such as vascular structure (vascularity (shape, clustered, uniform, non-clustered) presence of scale ( diffuse or in patches or grooves, etc.), orange structural areas or specific clues will be evaluated. If vascularity is detected at x200 magnification in patients undergoing lesional capillaroscopy, characterization of vascularity (point, clustered, uniform, etc.) will be made.

After dermoscopic criteria are determined, the individuals whose dermatology education range from 1 to 15 years will be randomized and divided into two groups, and the correct diagnosis rates will be measured, with one group only clinical and the other group clinical and dermoscopy images together.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have clinical/histopathological diagnosis of mycosis fungoides or parapsoriasis
* over the age of 18
* who have not received topical treatment for the last 2 weeks or systemic therapy for 4 weeks.
* patient who have patch lesions on their body

Exclusion Criteria:

* Patient who do not have clinical/histopathological diagnosis of mycosis fungoides or parapsoriasis
* under the age of 18
* who have received topical treatment for the last 2 weeks or systemic therapy for 4 weeks.
* patient who does not have patch lesions on their body

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were applied to Istanbul Teaching and Research hospital dermatology clinic between february 2022 and june 2022 and who meet each eligibility criteria were included to the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Correlation between videodermoscopy/capillaroscopy findings and histopathological findings of mycosis fungoides and parapsoriasis patients | 1 day (cross-sectional)
  Videodermoscopy/capillaroscopy and histopathological data will be recorded and evaluated for corelation

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Esra Koku Aksu, MD, Study Chair — Istanbul Teaching and Research Hospital
Locations (1):
- Istanbul Teaching and Research Hospital, Istanbul, Istanbul/Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lallas A, Apalla Z, Lefaki I, Tzellos T, Karatolias A, Sotiriou E, Lazaridou E, Ioannides D, Zalaudek I, Argenziano G. Dermoscopy of early stage mycosis fungoides. J Eur Acad Dermatol Venereol. 2013 May;27(5):617-21. doi: 10.1111/j.1468-3083.2012.04499.x. Epub 2012 Mar 9. PMID 22404051
- [Background] Xu C, Liu J, Wang T, Luo Y, Liu Y. Dermoscopic patterns of early-stage mycosis fungoides in a Chinese population. Clin Exp Dermatol. 2019 Mar;44(2):169-175. doi: 10.1111/ced.13680. Epub 2018 Jun 6. PMID 29876963